CLINICAL TRIAL: NCT06301841
Title: Prospective Randomized Clinical Trial Assessing the Value of an Antibiotic Protocol Guided by a Multimodal Approach in AECOPD With Pneumonia in Intensive Care
Brief Title: An Antibiotic Protocol Guided by a Multimodal Approach in AECOPD With Pneumonia in Intensive Care
Acronym: BPCTréa2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A00903-42
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: To Reduce Duration of Antibiotics Exposure in Patients With COPD Hospitalized in Intensive Care Unit With Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Conventional microbiological investigations are performed as soon as possible after ICU admission including blood cultures, non-invasive or invasive respiratory tract sample, urine antigen assays and viral PCR.
  Antibiotics have to be started as soon as possible after ICU admission and during at less 3 days
- Intervention (Experimental): In addition to conventional microbiological investigations, a non-invasive or invasive respiratory tract sample is collected as soon as possible and tested with the respiratory broad-panel mPCR (Biofire FilmArray Pneumonia plus Panel de Biomérieux). This test detects 18 bacteria, 9 viruses and 7 antibiotic resistance markers. In addition a procalcitonin assay is performed on day-3 of ICU admission.
  Antibiotics have to be started as soon as possible after ICU admission and during at less 3 days.
  At day 3, clinicians have to consider all the early microbiological results (including the respiratory broad-panel mPCR (Biofire FilmArray Pneumonia plus Panel de Biomérieux) and procalcitonin, and subsequently to apply an algorithm of early antibiotics discontinuation or de-escalation.
  Interventions: Other: experimental

INTERVENTIONS:
Other: experimental — At day 3, clinicians have to consider all the early microbiological results (including the respiratory broad-panel mPCR (Biofire FilmArray Pneumonia plus Panel de Biomérieux) and procalcitonin, and subsequently to apply an algorithm of early antibiotics discontinuation or de-escalation.
  Discontinuation is encouraged in case of no bacteria documentation and a procalcitonin < 1 ng/L; discontinuation is even encouraged if a viral documentation is concurrently obtained. In case of no bacteria documentation and a procalcitonin > 1 nd/L, antibiotic continuation is encouraged for additional two days.
  In case of bacteria documentation, antibiotic continuation is encouraged, but with narrowing the spectrum as much as possible. The duration of antibiotics is based on a procalcitonin algorithm: procalcitonin < 0.1 nd/l: discontinuation; 0.1 ng/l < procalcitonin < 0.25 ng/l: additional 1 day; procalcitonin > 0.25 ng/l: additional 2 days.
  Arms: Intervention

SUMMARY:
Investigators propose to conduct a multicenter, prospective, randomized, controlled, assessing the interests of an antibiotic protocol guided by the combined use of serum procalcitonin (PCT) and a broad-panel respiratory multiplex PCR (mPCR) to reduce duration of antibiotics exposure in patients with chronic obstructive pulmonary disease (COPD) hospitalized in intensive care unit (ICU) with pneumonia. The primary endpoint is the number of antibiotic-days for the treatment of pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Documented or suspected clinically COPD according to the criteria of GOLD
* Community-acquired pneumonia defined as the presence of a radiological (i.e., chest X-ray or CTscan) infiltrates consistent with an infectious site and associated with one or more of the following items: dyspnea, cough, sputum, fever above 38 ° C, chest pain, localized crackles with or without signs of pleural effusion, higher leukocytosis at 10,000 / mm³ or leukopenia below 4000 / mm³
* Admitted to the hospital for less than 48 hours
* ICU Admission
* Informed Consent signed by the patient or his representative

Exclusion Criteria:

* Patient immunocompromised including congenital immunodeficiency, haematologic malignancy, immunosuppressive drugs (including anticancer chemotherapy and post-transplantation therapies), neutropenia neutrophil count below 500 / mm³ secondary to chemotherapy, corticosteroids greater than 0.5 mg / kg / day for more than 10 days, HIV infection
* Therapeutic limitation Existence
* Minor patient or under guardianship or custody
* Pregnant woman
* Refusal to participate in the study
* The inclusion of the subject in another biomedical research protocol in progress or for less than 30 day
* Patients treated with antibiotics before ICU referral are no excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Duration of antibiotic therapy | from ICU admission to day 28 or hospital discharge
  The number of antibiotic-days for the treatment of pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: cedric daubin, MD, Principal Investigator — CHU de Caen Normandie, Médecine Intensive et Réanimation Médicale, 14000 CAEN, France
Locations (1):
- Medical Intensive Care Unit, CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: No